CLINICAL TRIAL: NCT01413451
Title: A Single-Dose Pilot Study of Radiolabeled Amatuximab (MORAb-009) in Mesothelin Over Expressing Cancers
Brief Title: Amatuximab for High Mesothelin Cancers
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110212; 11-C-0212
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-11-15

CONDITIONS: Carcinoma, Pancreatic Ductal; Mesothelioma; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Monoclonal IgG Antibody; Biodistribution; Pharmacokinetics; HACA; Safety; Mesothelioma; Ovarian Cancer; Pancreatic Duct Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Mesothelioma; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — amatuximab

INTERVENTIONS:
Drug: Amatuximab (MORab-009)

SUMMARY:
Background:

- Amatuximab is a cancer treatment drug that targets mesothelin. High levels of this substance are found on some kinds of tumor cells. Lab studies have shown that amatuximab helps the immune system to kill cells that have high levels of mesothelin. However, more research is needed to determine how safe and effective amatuximab is for treating tumors with high levels of mesothelin.

Objectives:

- To assess the safety and effectiveness of amatuximab in treating tumors with high levels of mesothelin.

Eligibility:

- Individuals at least 18 years of age who have a type of cancer that overexpresses mesothelin.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood tests and tumor assessment studies.
* Participants will have two intravenous doses of amatuximab several hours apart. Researchers will monitor them closely and do frequent blood draws. On the same day and also within 48 hours of the second dose, participants will have imaging studies. These studies will measure how well the amatuximab is working against the cancer.
* Participants will have a third imaging study of the cancer about 1 week after the infusions.
* Participants will have a followup visit 2 weeks after receiving amatuximab. This visit will require blood samples. Four weeks after receiving the drug, researchers will review patients symptoms or side effects. This interview can be done in person or by phone.

DETAILED DESCRIPTION:
Background:

* Amatuximab is a high-affinity monoclonal IgG antibody raised against human mesothelin.
* Mesothelin is a glycosyl-phosphatidyl inositol-linked membrane glycoprotein thought to be involved in tumor metastasis
* Mesothelin is over-expressed in many cancers

Objectives:

-The primary objective is to determine the biodistribution of radiolabeled amatuximab in tumor and nontumor tissues in subjects with mesothelin over-expressing cancers including mesothelioma, pancreatic, ovarian, and non small cell lung cancer.

Eligibility:

* Female or male subjects greater than or equal to 18 years of age;
* Histologically confirmed mesothelin-expressing cancer;
* Transaminases less than or equal to 3 times ULN for mesothelioma, non small cell lung and ovarian cancer;
* Transaminases less than or equal to 5 times ULN for pancreatic cancer with known liver metastasis.

Design:

* This is a single-center, single-dose, open-label, pilot study of MORAb-009 in approximately 20 subjects with mesothelin expressing tumors.
* Indium-radiolabeled MORAb-009 (5mCi) will be administered.
* Serial single photon emission-computerized tomography imaging will be performed to determine binding to tumor and nontumor tissue.
* Subjects will be observed closely for safety and possible development of anti-MORAb-009 antibodies.
* Pharmacokinetics of radiolabeled antibody will be determined with imaging over time.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Female or male subjects, greater than or equal to 18 years of age.
* Histologically-confirmed diagnosis of pancreatic adenocarcinoma, mesothelioma, mesothelin-positive ovarian cancer, or NSCLC. A new biopsy is not required; the diagnostic biopsy sample will be sufficient. IHC confirmation of mesothelin-positivity is not necessary for pancreatic adenocarcinoma and mesothelioma as nearly 100% of pancreatic adenocarcinomas and mesotheliomas express mesothelin. Mesothelin expression in ovarian cancer and NSCLC will be tested by IHC and any degree of positivity (1+, 2+, or 3+) will be accepted.
* Subjects are required to have measurable disease that has progressed through prior therapy and that includes a non-hepatic lesion for imaging that is greater than or equal to 1.5 cm, as defined by Modified Response Evaluation Criteria in Solid Tumors (RECIST).
* Eastern Cooperative Oncology Group (ECOG) performance status or 0, 1, or 2.
* Female subjects of childbearing potential and all male subjects are required to consent to use a medically acceptable method of contraception throughout the study period and for 30 days after amatuximab administration. A barrier method of contraception is required.
* Laboratory and clinical results within the 2 weeks prior to Day of Infusion as follows:

  * Absolute neutrophil count (ANC): greater than or equal to 1.5 times 10(9)/L
  * Platelet count: greater than or equal to 75 times 10(9)/L
  * Hemoglobin: greater than or equal to 9 g/dL
  * Serum bilirubin: less than or equal to 1.5 mg/dL
  * Aspartate transaminase (AST): less than or equal to 3 x upper limit of normal (ULN) (less than or equal to 5 ULN acceptable for pancreatic patients with known liver metastasis only)
  * Alanine transaminase (ALT) less than or equal to 3 times upper limit of normal (ULN) (less than or equal to 5 ULN acceptable for pancreatic patients with known liver metastasis only)
  * Alkaline Phosphatase less than or equal to 5 times ULN
  * Serum creatinine less than or equal to 1.5 mg/dL
* Subjects are required to be willing and able to provide written informed consent.

EXCLUSION CRITERIA:

* Subjects are ineligible to participate in this study if any of the following criteria are met:

  * Known allergy or hypersensitivity to monoclonal antibodies;
  * Prior treatment with amatuximab;
  * Prior treatment with SS1(dsFv)PE38 (SS1P);
  * Known brain metastases;
  * Known prosthetic devices that would prohibit imaging of lesion of interest due to radiographic artifact;
  * Evidence of other active malignancy requiring treatment;
  * Clinically significant heart disease (e.g., congestive heart failure of New York Heart Association Class III or IV, angina not well controlled by medication, or myocardial infarction within 6 months);
  * ECG demonstrating clinically significant arrhythmias. Subjects with chronic atrial arrhythmia, (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia), are eligible;
  * Active serious systemic disease, including active bacterial or fungal infection within 2 weeks before study entry;
  * Active viral hepatitis or symptomatic human immunodeficiency virus (HIV) infection;
  * Treatment within 3 months with immunomodulatory therapy (e.g., interferons, immunoglobulin therapy, Interleukin 1 receptor antagonist (IL-1RA) or systemic corticosteroids). Short-term systemic corticosteroids or topical or intra-articular steroids are acceptable, at the discretion of the Investigator;
  * Chemotherapy, biologic therapy, radiation therapy or immunotherapy within 3 weeks prior to dosing with amatuximab;
  * Breast-feeding, pregnant, or likely to become pregnant during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-07-12; Primary Completion 2013-11-15 (Actual); Study Completion 2013-11-15 (Actual)

PRIMARY OUTCOMES:
Biodistribution of radiolabelled amatuximab in tumor and nontumor tissues.
Tumor
Background ratio of maximum counts

SECONDARY OUTCOMES:
CTCAE V.4 events
Observation of HACA
PKs
Antibody uptake vs. IHC mesothelin expression

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hassan R, Ebel W, Routhier EL, Patel R, Kline JB, Zhang J, Chao Q, Jacob S, Turchin H, Gibbs L, Phillips MD, Mudali S, Iacobuzio-Donahue C, Jaffee EM, Moreno M, Pastan I, Sass PM, Nicolaides NC, Grasso L. Preclinical evaluation of MORAb-009, a chimeric antibody targeting tumor-associated mesothelin. Cancer Immun. 2007 Dec 19;7:20. PMID 18088084
- [Background] Hassan R, Ho M. Mesothelin targeted cancer immunotherapy. Eur J Cancer. 2008 Jan;44(1):46-53. doi: 10.1016/j.ejca.2007.08.028. Epub 2007 Oct 22. PMID 17945478
- [Background] Gubbels JA, Belisle J, Onda M, Rancourt C, Migneault M, Ho M, Bera TK, Connor J, Sathyanarayana BK, Lee B, Pastan I, Patankar MS. Mesothelin-MUC16 binding is a high affinity, N-glycan dependent interaction that facilitates peritoneal metastasis of ovarian tumors. Mol Cancer. 2006 Oct 26;5(1):50. doi: 10.1186/1476-4598-5-50. PMID 17067392